CLINICAL TRIAL: NCT00720031
Title: Treatment of Metastatic Melanoma With Autologous Melan-A/MART-1 Specific CTL Clones
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: general director, Nantes University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD 98/9-C
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2008-07

CONDITIONS: Immunotherapy
Keywords: Melanoma,; Melan-A tumor reactive T cell clones,; immunotherapy; HLA-A2 melanoma patients with; either loco-regional or lymphnode metastasis; transit nodules not surgically resectable; -measurable cutaneous or visceral metastasis .; Patients' tumor express Melan-A/MART-1 antigen.
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: autologous Melan-A/MART-1 specific CTL clones — By using patients' blood, several million to several billion of Melan-A/MART1 tumor reactive T cell clone(s) will be produced in vitro, then infused to the patient, 3 to 6 months after collecting blood sample. During this production period of the T cell clone, the patient will be treated with deticene at the dose of 250mg/m2/j by IV for 4 days each month.
  After each T cell clone infusion (J1), the patient will receive IFN-α at the dose of 9 M/U 3 times a week for 4 weeks and Interleukin-2 at the dose of 9 M/U from Day 1 to day 5 and from Day 8 to Day 12.

SUMMARY:
Most of HLA-A2 melanomas express Melan-A/MART-1 antigen and are recognized by tumor reactive Melan-A specific T lymphocytes. By using blood samples from HLA-A2 melanoma patients (stage III and IV), our goal is to produce a tumor reactive Melan-A specific T cell clones and to conduct a phase I-II clinical trial, based on the infusion of several millions to several billions of these lymphocytes to the patient, in order to induce passive immunity against this antigen. Production of the clones will be performed in the Unit for Cellular and Gene Therapy from Nantes University Hospital. Therapeutic response, safety treatment but also localization and survival of infused T cell clones will be assessed. This approach is expected to precise the ability of the clones to migrate within the tumor and to transfer specific immunity.

ELIGIBILITY:
Inclusion Criteria:

* HLA-A2 melanoma patients with :

  * either loco-regional or lymph node metastasis
  * transit nodules not surgically resectable
  * measurable cutaneous or visceral metastasis
* Patients' tumor express Melan-A/MART-1 antigen.
* No chemotherapy treatment (except for Deticene used before the first T cell clones infusion) or radiotherapy or immunotherapy in the last 4 weeks before infusion.
* No other melanoma treatment during the protocol.
* Life expectancy should be greater than 6 months.
* General state with Karnowsky greater than 80, ECOG = 0, 1 or 2.
* Patient should be negative for HIV and B and C hepatitis.
* Biological parameters at the beginning of the study: leucocytes ³ 2000 elements per mm3, hemoglobin ³ 10.5g/dl, platelets ³ 100 000 per mm3, phosphatases alcalines transaminases £ 1 time 1/2 compared to the normal.
* Signed informed consent

Exclusion Criteria:

* Cardio-vascular pathologies, evoluting and uncontrolled, (severe HTA), cardiac deficiency, severe angor, severe arrhythmia.
* Infectious pathologies evoluting and requiring antibiotherapy.
* Patients HIV+.
* Transplanted patients or patients suffering from severe auto-immune disease.
* Psychiatric troubles that do not allow the protocol follow-up.
* Pregnant or breast-feeding women.
* No contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2000-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of an adoptive immunotherapy specific for Melan-A/MART1 antigen in metastatic melanoma patients whose tumor express this antigen but also HLA-A2 | one year

SECONDARY OUTCOMES:
Evaluate whether infused T cell clones migrate to tumor sites. For this purpose, infused T cell clones will be characterized according to their Vß and Valpha using antibodies and/or PCR | after treatment
Evaluate whether infused T cell clones transfer a specific immunity. | J56 after treatment
evaluate infused Melan-A/MART1 reactive T cell clones tolerance | one year

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte DRENO, PhD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hopspital, Nantes, Pays de la Loire Region, France

REFERENCES:
- [Derived] Khammari A, Nguyen JM, Saint-Jean M, Knol AC, Pandolfino MC, Quereux G, Brocard A, Peuvrel L, Saiagh S, Bataille V, Limacher JM, Dreno B. Adoptive T cell therapy combined with intralesional administrations of TG1042 (adenovirus expressing interferon-gamma) in metastatic melanoma patients. Cancer Immunol Immunother. 2015 Jul;64(7):805-15. doi: 10.1007/s00262-015-1691-7. Epub 2015 Apr 7. PMID 25846669